CLINICAL TRIAL: NCT02625233
Title: Clinical Long-Term Evaluation of Approved and Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5788
Record Dates: First submitted 2015-11-03; First posted 2015-12-09 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Visual Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- senofilcon C (Experimental): Vistakon Investigational Contact Lens (Test)
  Interventions: Device: senofilcon C
- comfilcon A (Active Comparator): Marketed Monthly Wear Contact Lens (Control)
  Interventions: Device: comfilcon A

INTERVENTIONS:
Device: senofilcon C
  Arms: senofilcon C
Device: comfilcon A
  Arms: comfilcon A

SUMMARY:
This is a multi-site, dispensing, 4-visit, 2-arm parallel group, randomized, double-masked clinical trial using a Vistakon investigational contact lens (test) and a marketed monthly replacement contact lens (control). Each subject will be assigned randomly to either the test or control lens to evaluate the long term safety and efficacy of the investigational contact lens compared to the marketed contact lens over a period of six months of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 years of age.
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 in each eye.
* The subject's refractive cylinder must be ≤ 1.00 Diopters (D) in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.
* The subject should own a wearable pair of spectacles and bring to initial visit.
* The subject must be an adapted frequent replacement daily wear spherical silicone hydrogel soft contact lens wearer in both eyes.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* The subject must have enrolled and completed all visits in clinical study (NCT02515994).

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g., hepatitis, tuberculosis).
* Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g., Accutane), oral tetracyclines, topical scopolamine, oral phenothiazines (e.g. Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or OTC ocular medication.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any known hypersensitivity or allergic reaction to Opti-Free® PureMoist® multipurpose care solution or Eye-Cept rewetting drop solution
* Any ocular infection, allergy or clinically significant ocular disease (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Daily disposables, extended wear, monovision or multi-focal contact lens correction.
* History of binocular vision abnormality or strabismus.
* Employee or relative of employees of sponsor or investigational clinic (e.g., Investigator, Coordinator, Technician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vue Optical Boutique, Jacksonville, Florida
  - Omega Vision Center, PA / Sabal Eye Care, Longwood, Florida
  - Eyecare Associates, Bloomington, Illinois
  - Dr. Debbie H. Kim, OD, Closter, New Jersey
  - Sacco Eye Group, Vestal, New York
  - Dr. William Bogus, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 105 subjects were enrolled into this study. Of the enrolled subjects all were dispensed a study lens. Out of all the dispensed subjects 103 completed the study while 2 subjects were discontinued.
Groups:
- Senofilcon C: Subjects that wore the senofilcon C lens throughout the entire duration of the study.
- Comfilcon A: Subjects that wore the comfilcon A lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Senofilcon C | Comfilcon A
Started | 49 | 56
Completed | 47 | 56
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon C | Comfilcon A | Total
Number analyzed (Participants) | 49 | 56 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (7.03) | 31.5 (7.31) | 31.4 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 13 | 21 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3 | 3 | 6
  Black or African American | 3 | 1 | 4
  White | 43 | 52 | 95
Region of Enrollment [Number; unit: Participants]
  United States | 49 | 56 | 105

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes Grade 3 or Higher SLF
Description: Slit lamp findings were graded using a FDA Grade Scale, 0 = None, 1 = Slight, 2 = Moderate, 3 = Significant, 4 = Advanced. Measurements were taken in each subject eye at the initial visit, 4 month, 5 month and 6 month follow-up evaluations. This study is a continuation of a previous study therefore data from the initial visit was included in reporting. The proportion of subject eyes with SLF grade 3 or higher was reported for each lens.
Time Frame: Up to 6 Month Follow-up
Population: Subjects that were dispensed a study lens.
Measure: Number; unit: Proporiton of Subject Eyes
Units Other Than Participants: Subject Eyes
Groups:
- Senofilcon C: Subjects that wore the senofilcon C lens througout the entire duration of the study.
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 47 | 56
Number analyzed (Subject Eyes) | 376 | 448
Proporiton of Subject Eyes | 0 | 0

2. Primary Outcome: Visual Acuity (logMAR)
Description: The visual acuity (LogMAR) was collected at the initial visit, 4 month, 5 month and 6 month follow-up evaluations. This study is a continuation of a previous study therefore data from the initial visit was included in reporting. The average Visual Acuity (logMAR) across the 4 study visits and at each individual visit was reported for each lens.
Time Frame: Up to 6 Month Follow-up
Population: Subjects that completed all study visits.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Subject Eyes
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 47 | 56
Number analyzed (Subject Eyes) | 376 | 448
LogMAR
  Overall N=376, N=448 | -0.12 (0.066) | -0.12 (0.074)
  Initial Visit N=94, N=112 | -0.14 (0.069) | -0.13 (0.064)
  4 Month Follow-up N=94, N=112 | -0.12 (0.069) | -0.13 (0.075)
  5 Month Follow-up N=94, N=112 | -0.13 (0.068) | -0.12 (0.078)
  6 Month Follow-up N=94, N=112 | -0.12 (0.063) | -0.13 (0.072)

ADVERSE EVENTS:
Time Frame: Throught the duration of the study. Approximately 3 months per subject.
Description: NCT02625233 is a continuation of NCT02515994. Each study was approximately 3 months duration for each subject(i.e. if a subject was enrolled into both studies they wore the lens a total of 6 months). Refer to the adverse event information for study NCT02515994 for the previous 3 months.
Arm/Group | Senofilcon C | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/56
Other Adverse Events (participants affected / at risk) | 0/49 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days